CLINICAL TRIAL: NCT05617729
Title: A Clinical Simulation Study of a Test Material on the Anterior Nares
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Innovation and Research Organization (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Povinez001
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Colonization, Asymptomatic
MeSH Terms: conditions — Asymptomatic Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline (Placebo Comparator): this treatment consists of sterile saline that is applied to the nares using a swab
  Interventions: Other: Saline applied via swab
- Povidone-iodine based gel (Active Comparator): this treatment consists of a Povidone-Iodine based gel that is applied to the nares using a swab
  Interventions: Other: Povidone-iodine based gel

INTERVENTIONS:
Other: Saline applied via swab — sterile saline applied via swab
  Arms: Saline
Other: Povidone-iodine based gel — gel applied via swab
  Arms: Povidone-iodine based gel

SUMMARY:
The objective of this study is simulate the clinical use of a test material within a 24h window. Efficacy will be simulated as the capacity of the material to reduce or clear the anterior nares bacterial population from opportunistic pathogens (e.g. Staphylococcus Aureus, Escherichia Coli, etc).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female between 18 to 55 years of age;
2. Subject has normal nasal passage;
3. Subject has not history of chronic nasal passage disease (chronic rhinitis, chronic sinusitis).
4. Subject is willing to have materials applied and follow the protocol;
5. Subject agrees to avoid exposure of the test sites to any chemical product and to refrain from touching the area of application.
6. Subject agrees to refrain from getting the application site wet and scrubbing or washing the test area with soap or applying powders, lotions or personal care products to the area during the course of the study;
7. Subject agrees not to introduce any new cosmetic or toiletry products during the study;
8. Subject is dependable and able to follow directions as outlined in the protocol and anticipates being available for all study visits;
9. Subject is willing to participate in all study evaluations;
10. Subject is in generally good health;
11. Subject understands and is willing to sign an Informed Consent Form

Exclusion Criteria:

1. Female subject is pregnant, nursing, planning a pregnancy, or not using adequate birth control;
2. Subject has a chronic nasal disease (e.g sinusitis, rhinitis);
3. Subject has a bleeding disorder, immunologically compromised, recent illness/vaccination or currently febrile;
4. Subject reports a history of allergies to antiseptics;
5. Subject is currently taking certain medications which, in the opinion of the Principal Investigator, may interfere with the study;
6. Subject has known allergies to skin treatment products or cosmetics, toiletries, and/or topical drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Colony Forming Units | up to 24 hours following application

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Innovation and Research Organization, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Fernandez-Rodriguez D, Cho J, Chisari E, Citardi MJ, Parvizi J. Nasal microbiome and the effect of nasal decolonization with a novel povidone-iodine antiseptic solution: a prospective and randomized clinical trial. Sci Rep. 2024 Jul 20;14(1):16739. doi: 10.1038/s41598-023-46792-8. PMID 39033201